CLINICAL TRIAL: NCT00608556
Title: Ciliary Dysfunction as an Underlying Etiology Linking Primary Ciliary Dyskinesia With Heterotaxy and Complex Congenital Heart Disease
Brief Title: Dyskinesia, Heterotaxy and Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080067; 08-I-0067
Record Dates: First submitted 2008-02-04; First posted 2008-02-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-10-31

CONDITIONS: Ciliary Dyskinesia, Primary; Kartagener Syndrome; Congenital Heart Defects; Situs Inversus
Keywords: Heterotaxy; Primary Ciliary Dyskinesia; Congenital Heart Disease; Genetic Study; Situs Inversus
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome; Heart Defects, Congenital; Situs Inversus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine genetic material obtained from blood and tissue samples of patients with congenital heart disease (CHD) and heterotaxy (an abnormality in the left-right positioning of organs in the body, also called situs inversus) to gain a better understanding of these disorders and of a lung disease called primary ciliary dyskinesia (PCD). CHD is prevalent in patients with heterotaxy. It is believed that certain forms of CHD or heterotaxy may have the same genetic origin as PCD.

Individuals 2 years of age or older who have a CHD or heterotaxy or both may be eligible for this study. Participants undergo some or all of the following tests and procedures:

* Blood tests, electrocardiogram (EGC) and chest x-ray.
* Saliva collection: Subjects rinse their mouth with water, and then spit approximately 1.5 cc of saliva into a sterile container.
* Buccal swabs: A small soft, toothbrush-like swab is rubbed on the inside lining of the cheek to collect tissue samples.
* Nasal tests to measure nasal nitric oxide levels and to obtain tissue samples from the inside of the nostrils: For the nitric oxide level test, a rubber probe is inserted into one of the nostrils until it fits snugly and comfortably. The subject then takes a deep breath and then exhales all the way out through the mouth through a plastic device. During exhalation, gas measurements are recorded on a computer. To obtain tissue samples, a device is inserted in a nostril and scraped gently against the inside of the nose.
* Echocardiography: This ultrasound test of the heart uses sound waves to obtain pictures of the heart. A small wand with a warm clear gel is moved around the chest to obtain the images.
* Abdominal ultrasound: This ultrasound test of the heart uses sound waves to obtain pictures of the abdominal organs. A small wand with a warm clear gel is moved around the abdomen to obtain the images....

DETAILED DESCRIPTION:
The goal of this study is to elucidate the possible role of primary ciliary dyskinesia (PCD) in complex congenital heart disease associated with heterotaxy. This study arises from our recent finding of an unexpectedly high incidence (40 percent) of complex congenital heart disease together with heterotaxy in a mutant mouse model of PCD. These findings suggest heterotaxy can arise from mutations causing PCD. Consistent with this, a recent clinical research study showed some patients with PCD have undiagnosed heterotaxy. However, there has not been any clinical study to ascertain if patients diagnosed with heterotaxy may suffer from PCD, the focus of this IRB protocol. These studies are of immediate clinical importance, as heterotaxy patients undergoing surgical correction for complex structural heart defects can become ventilator dependent for unknown causes. A diagnosis of PCD in patients with heterotaxy would significantly alter clinical management strategies that have the potential to significantly improve outcome for heterotaxy patients undergoing high-risk cardiac surgery for complex congenital heart defects.

For this study, we will recruit pediatric subjects undergoing surgery for complex congenital heart defects associated with heterotaxy at Children's National Medical Center. We will also recruit adult patients with heterotaxy heart disease or situs inversus from the Children's National Medical Center and at NIH. In addition, we will recruit patients, ages 2 years and older, seen at the NIH by Dr. Kenneth Olivier with known PCD or Kartagener syndrome and with documentation or high clinical suspicion of heterotaxy or situs inversus into our study. Subjects will be evaluated for PCD using standard operating procedures (SOPs). This will include obtaining airway epithelial tissue samples to assess ciliary motion by videomicroscopy and for assessing defects in ciliary ultrastructure by electron microscopy. In addition, nasal nitric oxide measurements will be obtained, as reduced NO levels are often associated with PCD. All of these procedures will utilize SOPs obtained from approved IRB protocols that are part of a multi-center study at the University of North Carolina (Dr. Michael Knowles) and at the NIH (Dr. Ken Olivier, NIAID). In addition, blood, buccal swab, and saliva samples will be obtained for DNA analysis of candidate genes known to cause heterotaxy and/or PCD. Through these studies, we hope to establish whether mutations causing PCD may contribute to heterotaxy and situs anomalies. Such findings may suggest changes in the standard of care for heterotaxy patients to include the evaluation for PCD, particularly prior to surgery. In addition, the DNA analysis may provide novel insights into the genetic causes for complex congenital heart defects associated with heterotaxy and PCD, allowing the future development of appropriate diagnostic tests for more accurate identification of patients at risk for PCD. Together, the outcome of this study can have significant impact on improving the clinical care for patients with congenital heart disease associated with situs anomalies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients who have diagnosed congenital heart disease, heterotaxy or situs inversus will be asked to participate in this study regardless of sex, age, or race. In addition, patients who have diagnosed PCD or Kartagener syndrome with documentation or high clinical suspicion of heterotaxy or situs inversus will also be recruited to participate in this study. There is no known ethnic or racial predilection for heterotaxy, congenital heart disease, situs inversus, PCD, or Kartagener syndrome.

EXCLUSION CRITERIA:

Certain conditions may preclude specific procedures included in this protocol, but may still allow pertinent parts of the diagnostic evaluation. These conditions/procedures may include: pregnancy/chest radiograph. For reversible conditions, such as acute upper airway infection, significant epistaxis within the prior week (not related to number 2 below), or lower airway infection with uncontrollable coughing, the participant may need to be re-evaluated after resolution. For nasal NO or nasal mucosal scrapings, the following lists the absolute contraindications:

1. Anatomic abnormality of the nose or sinuses (e.g. complete sinus blockage or turbinatectomy) that precludes the measurement of nasal NO.
2. A severe bleeding diathesis or condition, such as hereditary hemorrhagic telangiectasia syndrome, that may predispose to significant nasal bleeding or result in a severely excoriated nasal mucosa.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-01-25; Study Completion 2011-10-31

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Aylsworth AS. Clinical aspects of defects in the determination of laterality. Am J Med Genet. 2001 Jul 15;101(4):345-55. PMID 11471158
- [Background] Bartoloni L, Blouin JL, Pan Y, Gehrig C, Maiti AK, Scamuffa N, Rossier C, Jorissen M, Armengot M, Meeks M, Mitchison HM, Chung EM, Delozier-Blanchet CD, Craigen WJ, Antonarakis SE. Mutations in the DNAH11 (axonemal heavy chain dynein type 11) gene cause one form of situs inversus totalis and most likely primary ciliary dyskinesia. Proc Natl Acad Sci U S A. 2002 Aug 6;99(16):10282-6. doi: 10.1073/pnas.152337699. Epub 2002 Jul 25. PMID 12142464
- [Background] Bisgrove BW, Yost HJ. The roles of cilia in developmental disorders and disease. Development. 2006 Nov;133(21):4131-43. doi: 10.1242/dev.02595. Epub 2006 Oct 4. PMID 17021045